CLINICAL TRIAL: NCT00218270
Title: Treatment of Smokeless Tobacco Users
Brief Title: Effectiveness of Using Tobacco Free Snuff in Reducing Negative Effects of Smokeless Tobacco Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Dorohty Hatsukami, UMN
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-14404-2; R01-14404-2; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2008-06

CONDITIONS: Tobacco Use Disorder
Keywords: Smokeless tobacco, harm reduction
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Reduction of tobacco use by substituting tobacco free snuff.
  Interventions: Drug: Tobacco free snuff
- 2 (Placebo Comparator): Reduction of tobacco use by using behavioral techniques.
  Interventions: Drug: Tobacco free snuff

INTERVENTIONS:
Drug: Tobacco free snuff — Tobacco free snuff
  Other Names: Smokey Mountain

SUMMARY:
Though spit tobacco is smokeless, it still affects the cardiovascular system and may be associated with heart disease, stroke, and high blood pressure. Long-term effects of smokeless tobacco (ST) include tooth abrasion, gum recession, mouth disease, loss of bone in the jaw, yellowing of teeth, and chronic bad breath. This study will assess the effectiveness of using tobacco free snuff in reducing levels of exposure to tobacco and associated toxicity, as well as enhancing motivation to either quit or sustain lower levels of nicotine intake.

DETAILED DESCRIPTION:
Spit tobacco presents as many health risks to its users as smoking tobacco. Although a significant number of ST users recognize the importance of quitting, many either do not want to quit or feel it is impossible. For these individuals, tobacco reduction may be an important transitional goal, either prior to quitting or as a treatment endpoint. However, approaches to help ST users reach this goal have not been studied. This study will assess the effectiveness of using tobacco-free snuff in reducing levels of exposure to tobacco and associated toxicity, as well as enhancing motivation to either quit or sustain lower levels of nicotine intake.

Participants will be randomly assigned to receive either treatment with tobacco-free snuff or treatment without it. All participants will be encouraged to reduce nicotine intake by 50% during the first four weeks and by 75% the following four weeks. Participants receiving the tobacco-free snuff will be asked to alternate the use of their usual brand of ST with tobacco-free snuff in order to achieve the targeted reduction. Participants not receiving the tobacco-free snuff will only be informed to try to cut down their tobacco use to the targeted reduction. Study visits will occur once weekly during the 8-week treatment period. Assessments will include vital signs, physiological measures related to tobacco use, and measures of motivation and self-efficacy to quit ST. The number of participants who either do not complete treatment, reduce nicotine intake, or quit completely will be assessed at the Week 8 study visit and at follow-up visits, which will be held at Weeks 12 and 26.

ELIGIBILITY:
Inclusion Criteria:

* Not interested in quitting smokeless tobacco use within 90 days of study entry
* Used smokeless tobacco at least six times a day for 6 months prior to study entry
* Agree to use an effective form of contraception throughout the study

Exclusion Criteria:

* Current use of tobacco or nicotine products other than ST
* Pregnant or breastfeeding
* Any unstable medical condition
* Use of any medication that may affect tobacco use or be affected by reduction of tobacco use
* DSM-IV diagnosis of any psychiatric disorders or substance abuse disorders within 6 months prior to study entry
* Use of any psychotropic medications within 6 months prior to study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2002-12; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Percent reduction in use | Week 8, 12, and 26
Toxicity profile of carcinogen metabolites | Week 8, 12, and 26
Number of unsuccessful quit attempts | Week 8, 12, and 26
Abstinence (measured at Weeks 8, 12, and 26) | Week 8, 12, and 26

SECONDARY OUTCOMES:
Motivation and self-efficacy (measured at Weeks 8, 12, and 26) | Week 8, 12, and 26

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States